CLINICAL TRIAL: NCT02670356
Title: Study Comparing Fish Oil and Krill Oil
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped by the company funding the study
Sponsor: Tufts University (Other)
Collaborators: Prevention Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Stefania lamon-Fava, Scientist I. Associate Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11787
Record Dates: First submitted 2015-12-23; First posted 2016-02-01 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Inflammation; Dyslipidemia
Keywords: fish oil; EPA; DHA; krill oil; Metabolic Syndrome
MeSH Terms: conditions — Inflammation; Dyslipidemias; Metabolic Syndrome | interventions — Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish oil (Experimental): fish oil, 1500 mg/day, EPA:DHA ratio of 4:1, each capsule containing 750 mg total EPA+DHA, 2 capsules/day for 10 weeks
  Interventions: Dietary Supplement: Fish oil
- krill oil (Experimental): krill oil, 300 mg/day, each capsule containing 74 mg total EPA+DHA , 1 capsule/day for 10 weeks
  Interventions: Dietary Supplement: Krill oil

INTERVENTIONS:
Dietary Supplement: Fish oil — two 750 mg/capsules/day
  Arms: Fish oil
Dietary Supplement: Krill oil — one 300 mg capsule/day
  Arms: krill oil

SUMMARY:
Eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are omega-3 fatty acids found in fish oil and in krill oil. The purpose of this study is to compare the effects of the recommended dose of a fish oil supplement (Omax3 4:1 EPA:DHA; recommended daily dose 1650 mg - totaling 1500 mg EPA+DHA) and a krill oil supplement (MegaRed; recommended daily dose 300 mg - totaling 74 mg EPA+DHA) on omega-3 index, plasma biomarkers of inflammation and inflammatory cell activation, and plasma lipid levels in subjects with metabolic syndrome.

DETAILED DESCRIPTION:
Inflammation plays a pivotal role in the pathogenesis of several chronic diseases including cardiovascular disease and diabetes mellitus. There has been some evidence that fish oil, containing the omega-3 fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), reduces the risk or severity of these diseases, leading several government and health organizations to advocate an increased consumption of fish or fish oil. Fish oil contains EPA and DHA either as triglycerides or as ethyl esters. Recently, krill oil has gained popularity as an EPA and DHA supplement. Krill oil contains EPA and DHA in phospholipid, triglyceride, and free fatty acid form.

Some studies have shown that the bioavailability of EPA and DHA in krill oil is higher than in fish oil and that smaller doses of krill oil are therefore sufficient to observe a significant effect on the desired outcome (inflammation, plasma lipid levels).

The central hypothesis of this proposal is that the dose of the EPA and DHA omega-3 fatty acids is more important than their bioavailability in effecting changes in systemic inflammation and lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* fasting plasma triglyceride levels between 150 and 500 mg/dL
* C-reactive protein (CRP) levels ≥2 µg/mL
* at least one of the following criteria for the definition of metabolic syndrome: abdominal obesity (waist circumference >40 inches in men and >35 inches in women), hypertension (blood pressure ≥130/≥85 mmHg or use of anti-hypertensive medications), and fasting glucose ≥110 mg/dL.

Exclusion Criteria:

* high-fish diets (>2 fish meals/week)
* taking fish oil supplements or supplements containing EPA or DHA
* regular use of anti-inflammatory medications
* Above normal coagulation time or use of anticoagulant medications
* allergy to fish, fish oil, or shellfish
* uncontrolled thyroid dysfunction
* insulin-dependent type 2 diabetes mellitus
* kidney or liver disease
* smoking
* drinking more than 7 alcoholic drinks/week
* use of lipid-lowering medications or medications known to alter lipoprotein metabolism

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Omega-3 index | 10 weeks
  red blood cell membrane levels of EPA and DHA, as percent of total fatty acids

SECONDARY OUTCOMES:
interleukin-6 (IL-6) | 10 weeks
  plasma levels as pg/mL
Tumor necrosis factor alpha (TNF-alpha) | 10 weeks
  plasma levels as pg/mL
Monocyte chemoattractant protein 1 (MCP-1) | 10 weeks
  plasma levels as pg/mL
Total cholesterol | 10 weeks
  plasma levels as mg/dL
LDL cholesterol | 10 weeks
  plasma levels as mg/dL
HDL cholesterol | 10 weeks
  plasma levels as mg/dL
TG | 10 weeks
  plasma levels as mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Lamon-Fava, Ph.D., Principal Investigator — Tufts University
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No